CLINICAL TRIAL: NCT06373900
Title: Wound Closure After Total Knee Arthroplasty: Comparison of Polypropylene and Polyglactin 910 Suture. A Randomised Controlled Trial.
Brief Title: Wound Closure After Total Knee Arthroplasty: Comparison of Polypropylene and Polyglactin 910 Suture.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indus Hospital and Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IndusH
Record Dates: First submitted 2024-03-25; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Wound Heal; Wound Dehiscence; Wound Complication

STUDY DESIGN:
Who Masked: Participant
Masking Description: SNOS protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): wound closure with polypropylene
  Interventions: Procedure: wound closure
- Group B (Active Comparator): wound closure with polyglactin 910 suture
  Interventions: Procedure: wound closure

INTERVENTIONS:
Procedure: wound closure — Group A wound will be closed with Polypropylene and Group B wound will be closed with Polyglactin 910 suture. both wound closure followed for healing, infection and scar formation till 30th post operative day.

SUMMARY:
Comparison of wound complication and scar formation in patient undergone bilateral total knee replacement comparison between polypropylene and polyglactin 910 suture. patient randomised according to SNOS protocol into group A and B for their right and left knee closure with each suture. patient followed on 3rd, 7th, 15th and 30th post operative day for wound healing, wound dehiscence and scar formation.

DETAILED DESCRIPTION:
All patients aged 50-80 years, belonging to either sex, diagnosed with end-stage osteoarthritis or post-traumatic arthritis, and scheduled for bilateral primary total knee arthroplasty at the Department of Orthopedics, Indus Hospital and Health Network, Karachi were enrolled in the study. Exclusion criteria included patients having existing skin, neuromuscular, or connective tissue disorders, rheumatoid arthritis, immunosuppression, morbid obesity, and pregnancy. All patients provided voluntary informed written consent before enrolment in the study.

In all patients undergoing primary TKA, one knee was closed using polypropylene, whereas the other was closed with Polyglactin 910 sutures. All surgeries were performed by the same surgical team using a standard medial parapatellar approach. The number of sutures and wound closure techniques were standardized across both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 to 80 years
* Both gender
* Inform consent
* End stage osteoarthritis

Exclusion Criteria:

* Age less the 50 and more then 80
* BMI more then 40
* Rheumatoid Arthritis
* lack of consent
* Pregnant female

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-13 (Actual); Primary Completion 2022-02-19 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Wound characteristics and complications | 30 days after surgery
  Post operative patient followed on 3rd, 7th, 15th and 30th day for the assessment of any erythema, wound dehiscence, discharge, blister around the wound, warmth and tenderness
Wound Infection Grade | 30 days after surgery
  wound infection grade assessed on post operative day 3rd, 7th, 15th and 30th as simple stitch abscess, surrounding cellulitis, any systematic symptoms or suture removed.
Hollander Cosmetic Wound Evaluation Score | 30 days after surgery
  Hollander score assessed on 3rd, 7th, 15th and 30th post operative day as step off border, contour, scar width, scar width, edge inversion and overall cosmesis

CONTACTS AND LOCATIONS:
Overall Officials: Nek Mohammad, Principal Investigator — The Indus Hospital and Health Network
Locations (1):
- Indus Hospital and Health Network, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khan MA, Memon MW, Chinoy A, Javed S, Barkat R, Jiwani A. Wound closure after total knee replacement: Comparison between staples and sutures. Pak J Med Sci. 2022 Jan;38(2):340-344. doi: 10.12669/pjms.38.ICON-2022.5782. PMID 35310806
- [Result] Li JW, Ma YS, Xiao LK. Postoperative Pain Management in Total Knee Arthroplasty. Orthop Surg. 2019 Oct;11(5):755-761. doi: 10.1111/os.12535. PMID 31663286
- [Result] Culliford D, Maskell J, Judge A, Cooper C, Prieto-Alhambra D, Arden NK; COASt Study Group. Future projections of total hip and knee arthroplasty in the UK: results from the UK Clinical Practice Research Datalink. Osteoarthritis Cartilage. 2015 Apr;23(4):594-600. doi: 10.1016/j.joca.2014.12.022. Epub 2015 Jan 9. PMID 25579802
- [Result] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Result] Maradit Kremers H, Visscher SL, Moriarty JP, Reinalda MS, Kremers WK, Naessens JM, Lewallen DG. Determinants of direct medical costs in primary and revision total knee arthroplasty. Clin Orthop Relat Res. 2013 Jan;471(1):206-14. doi: 10.1007/s11999-012-2508-z. PMID 22864619
- [Result] Faour M, Sodhi N, Khlopas A, Piuzzi NS, Stearns KL, Krebs VE, Higuera CA, Mont MA. Knee Position during Surgical Wound Closure in Total Knee Arthroplasty: A Review. J Knee Surg. 2018 Jan;31(1):6-12. doi: 10.1055/s-0037-1608838. Epub 2017 Nov 22. PMID 29166680
- [Result] Tajirian AL, Goldberg DJ. A review of sutures and other skin closure materials. J Cosmet Laser Ther. 2010 Dec;12(6):296-302. doi: 10.3109/14764172.2010.538413. PMID 21142740
- [Result] Agarwala S, Vijayvargiya M. Concealed cosmetic closure in total knee replacement surgery - A prospective audit assessing appearance and patient satisfaction. J Clin Orthop Trauma. 2019 Jan-Feb;10(1):111-116. doi: 10.1016/j.jcot.2017.11.002. Epub 2017 Nov 13. PMID 30705543
- [Result] Khan RJ, Fick D, Yao F, Tang K, Hurworth M, Nivbrant B, Wood D. A comparison of three methods of wound closure following arthroplasty: a prospective, randomised, controlled trial. J Bone Joint Surg Br. 2006 Feb;88(2):238-42. doi: 10.1302/0301-620X.88B2.16923. PMID 16434531
- [Result] Liu S, Wang Y, Kotian RN, Li H, Mi Y, Zhang Y, He X. Comparison of Nonabsorbable and Absorbable Suture in Total Knee Arthroplasty. Med Sci Monit. 2018 Oct 23;24:7563-7569. doi: 10.12659/MSM.910785. PMID 30350827
- [Result] Elbardesy H, Gul R, Guerin S. Subcuticular sutures versus staples for skin closure after primary hip arthroplasty. Acta Orthop Belg. 2021 Mar;87(1):55-64. PMID 34129758
- [Result] Newman JT, Morgan SJ, Resende GV, Williams AE, Hammerberg EM, Dayton MR. Modality of wound closure after total knee replacement: are staples as safe as sutures? A retrospective study of 181 patients. Patient Saf Surg. 2011 Oct 19;5(1):26. doi: 10.1186/1754-9493-5-26. PMID 22011354
- [Result] Yuenyongviwat V, Iamthanaporn K, Hongnaparak T, Tangtrakulwanich B. A randomised controlled trial comparing skin closure in total knee arthroplasty in the same knee: nylon sutures versus skin staples. Bone Joint Res. 2016 May;5(5):185-90. doi: 10.1302/2046-3758.55.2000629. PMID 27190132
- [Result] Hollander JE, Singer AJ, Valentine S, Henry MC. Wound registry: development and validation. Ann Emerg Med. 1995 May;25(5):675-85. doi: 10.1016/s0196-0644(95)70183-4. PMID 7741347
- [Result] Wyles CC, Jacobson SR, Houdek MT, Larson DR, Taunton MJ, Sim FH, Sierra RJ, Trousdale RT. The Chitranjan Ranawat Award: Running Subcuticular Closure Enables the Most Robust Perfusion After TKA: A Randomized Clinical Trial. Clin Orthop Relat Res. 2016 Jan;474(1):47-56. doi: 10.1007/s11999-015-4209-x. PMID 25733009

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT06373900/Prot_SAP_ICF_000.pdf